CLINICAL TRIAL: NCT06405113
Title: Fecal Microbiota Transplantation Combined with SOX and Sintilimab As First-line Treatment for Advanced Gastric Cancer:A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Study (FMT-JSNO-01)
Brief Title: FMT+SOX+Sintilimab As First-line Treatment for Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Hua Jiang, MD, Changzhou No.2 People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: [2024]YLJSA001
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Fecal Microbiota Transplantation(FMT)+SOX+Sintilimab
  Interventions: Combination Product: Fecal Microbiota Transplantation (FMT)+chemotherapy+immunotherapy
- Placebo Comparator Arm (Placebo Comparator): Placebo+SOX+Sintilimab
  Interventions: Combination Product: Fecal Microbiota Transplantation (FMT)+chemotherapy+immunotherapy

INTERVENTIONS:
Combination Product: Fecal Microbiota Transplantation (FMT)+chemotherapy+immunotherapy — Participants received Fecal Microbiota Transplantation (FMT) combined with (Oxaliplatin + S-1)+Sintilimab

SUMMARY:
the investigators plan to initiate a prospective, multicenter, randomized, double-blind, placebo-controlled phase II study, recruiting 198 patients with advanced gastric/gastroesophageal junction adenocarcinoma who have not received prior treatment. Randomly divided into two groups, one group is the group of fecal microbiota transplantation(FMT)+SOX+Sintilimab, and the other group is the group of SOX+Sintilimab. Compare the 2-year OS rates of the two groups to verify whether the addition of FMT to first-line treatment can improve the prognosis of gastric cancer patients.

DETAILED DESCRIPTION:
the investigatorse plan to initiate a prospective, multicenter randomized, double-blind, placebo-controlled phase II study, recruiting a total of 198 patients with previously untreated unresectable advanced or metastatic gastric/gastroesophageal junction adenocarcinoma in our hospital and 14 other hospitals. Randomly divided into Group A and Group B, Group A received FMT+SOX chemotherapy regimen +Sintilimab immunotherapy regimen, Group B only received SOX chemotherapy regimen+and Sintilimab immunotherapy regimen. If there is no progression of the disease after 4-6 cycles of first-line treatment, both groups of patients will enter the first-line maintenance treatment stage: S-1+Sintilimab, until disease progression, intolerance, or death occurs. The aim is to explore the efficacy and safety of FMT combined with SOX and Sintilimab in the treatment of advanced first-line gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-80 (including 18 and 80 years old);
* Understand the research steps and content, and voluntarily sign a written informed consent form;
* Non resectable Her-2 negative advanced or metastatic gastric/gastroesophageal junction adenocarcinoma confirmed by histopathology and/or cytology, excluding all other histological types;
* At least one measurable lesion, according to RECIST 1.1 standard;
* Have not received anti-tumor treatment in the past;
* The physical status score of Eastern Tumor Collaboration Group (ECOG) was 0-1;
* Expected survival time ≥ 3 months;
* Have adequate organ and bone marrow function, laboratory examination within 7 days prior to enrollment meets the following requirements (no blood components, cell growth factors, albumin or other corrective drugs are allowed within 14 days prior to obtaining laboratory examination), as follows: 1) Blood routine: absolute neutrophil count (ANC) ≥1.5×109/L, platelet (PLT) ≥75×109/L, hemoglobin (HGB) ≥90 g/L (no blood transfusion or erythropoietin dependence within 14 days); 2) Liver function: serum total bilirubin (TBIL) ≤2 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 5x ULN, serum albumin ≥28 g/L; alkaline phosphatase (ALP) ≤5×ULN; 3) Renal function: serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥50 mL/min (using the standard Cockcroft-Gault formula) : Urine routine results showed urinary protein < 2+; For patients with urine protein ≥2+ at baseline,24-hour urine collection and 24-hour urine protein quantification<1g should be performed; 4) Coagulation function: International standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN; If the subject is receiving anticoagulant therapy, as long as the INR is within the intended range of anticoagulant drug use.
* For female subjects of reproductive age, a urine or serum pregnancy test should be performed and the result is negative 3 days prior to receiving the initial study drug administration;
* Subjects and their sexual partners are required to use a medically approved contraceptive method (such as an IUD, contraceptive pill, or condom) during the study treatment period and for 6 months after the end of the study treatment period.

Exclusion Criteria:

* Currently participating in an interventional clinical study or receiving another investigational drug or investigational device within 4 weeks prior to initial dosing;
* Received proprietary Chinese medicines with anti-tumor indications or immunomodulatory drugs (thymosin, interferon, interleukin, etc.) within 2 weeks before the first administration, or received major surgical treatment within 3 weeks before the first administration;
* Class III - IV congestive heart failure (New York Heart Association classification), poorly controlled and clinically significant arrhythmias;
* Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before treatment;
* Known allergic reaction to the drug in this study;
* Patients requiring long-term systemic use of corticosteroids. Patients with COPD or asthma requiring intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroids could be enrolled;
* Symptomatic central nervous metastases. Patients with asymptomatic BMS or BMS whose symptoms are stable after treatment are eligible to participate in this study if they meet all of the following criteria: measurable lesions outside the central nervous system; No midbrain, pontine, cerebellum, meninges, medulla oblongata or spinal cord metastasis; Maintain clinical stability for at least 2 weeks;
* Stop hormone therapy 3 days before the first dose of the study drug;
* There is an active infection requiring treatment or systemic anti-infective drugs have been used in the week prior to the first dosing;
* Has not fully recovered from toxicity and/or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or baseline, excluding weakness or hair loss);
* Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
* Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greater than the upper limit of normal value in the laboratory of the study center);
* Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
* Pregnant or lactating women;
* Medical history or evidence of disease that may interfere with test results, prevent participants from fully participating in the study, abnormal treatment or laboratory test values, or other conditions that the investigator considers unsuitable for enrollment The Investigator considers other potential risks unsuitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival rate(2year-OS Rate) | up to 24 months
  The proportion of patients who have not died after 2 years of treatment

SECONDARY OUTCOMES:
Median Progression-Free Survival (mPFS) | up to 24 months
  Observation for mPFS will be recorded until the end of follow-up after the start of 1st cycle of treatment.
Objective Response Rate (ORR) | up to 24 months
  Objective response rate will be assessed by investigators.
Incidence of Adverse events (AEs) | up to 24 months
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
The Diversity of Fecal Microbiota | up to 24 months
  This will be detected by 16s rRNA sequencing or metagenomes.
Quality of Life (QoL) | up to 24 months
  QoL will be evaluated by EORTC-QLQ-C30.

CONTACTS AND LOCATIONS:
Locations (1):
- Changzhou No.2 People's Hospital, Changzhou, China

IPD SHARING:
Plan to Share IPD: No